CLINICAL TRIAL: NCT05247424
Title: Pretreatment With Unfractionated Heparin for ST Elevation Myocardial Infarction
Acronym: UFH-STEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Peter Radsel, Head of intensive internal medicine department, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Heparin-STEMI
Record Dates: First submitted 2022-01-30; First posted 2022-02-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: Myocardial Reperfusion; Unfractionated heparin; pre-treatment
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: randomization in 1:1 ratio
Who Masked: Outcomes Assessor
Masking Description: Interventional cardiologists evaluating coronary angiography will be blinded to assigned group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early unfractionated heparin (Experimental): Administration of UFH at a dose of 100 IU/kg body weight at first medical contact. Addition of UFH before coronary intervention according to ACT measurement after coronary angiography before coronary intervention.
  Interventions: Drug: Unfractionated heparin
- Control - Unfractionated heparin for coronary intervention only (No Intervention): Control arm with administration of UFH at a dose of 100 IU/kg body weight after coronary angiography before coronary intervention.

INTERVENTIONS:
Drug: Unfractionated heparin — Unfractionated heparin at dose of 100 IU /kg body weight
  Arms: Early unfractionated heparin

SUMMARY:
Rupture of a coronary artery plaque leads to thrombotic occlusion of the coronary artery and would present as ST segment elevation myocardial infarction. Early treatment with aspirin and early primary percutaneous coronary intervention are indicated. Anticoagulation therapy, usually with unfractionated heparin, is required during percutaneous coronary intervention.

Investigators hypothesis is that pretreatment with unfractionated heparin in addition to aspirin at first medical contact may facilitate spontaneous reperfusion of culprit artery and procedural thrombotic complication in patients with ST elevation myocardial infarction without significant risk of bleeding complications.

DETAILED DESCRIPTION:
Randomization of patients with STEMI at first medical contact in a 1:1 ratio into an intervention group receiving 100 IU of unfractionated heparin (UFH) per kilogram of body weight IV and later additionally UFH after diagnostic coronary angiography according to the activated clotting time (ACT) and a control group receiving only UFH after diagnostic coronary angiography at the dose of 100 IU per kilogram of body weight.

The primary end point of the study is TIMI flow at coronary angiography. Secondary endpoints are: Bleeding complications (defined by BARC score), occurrence of cardiogenic shock, and 30-day mortality.

Investigators plan to randomize 600 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with STEMI referred for primary PCI
* Duration of symptoms less than 6 hours before presentation

Exclusion Criteria:

* Pregnancy
* Cardiogenic shock at presentation (hemodynamic instability)
* Cardiac arrest before randomization
* Duration of symptoms for more than 6 hours before presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
TIMI flow | Day 0
  TIMI flow in culprit coronary artery at first coronary angiography

SECONDARY OUTCOMES:
Bleeding | Day 0
  Bleeding assessed by Bleeding Academic Research Consortium (BARC) score. BARC incorporates 5 bleeding types, ranging from BARC 0 - no bleeding to BARC 5 - fatal bleeding.
Cardiogenic shock | Day 0 to 10
  Presence of cardiogenic shock at any time after randomization
30 day mortality after STEMI | 30 days
  30-day mortality after STEMI
Troponin I concentration 24 h after primary PCI | 24 h
  Troponin I concentration 24 h after primary PCI

CONTACTS AND LOCATIONS:
Overall Officials: Miša Fister, MD, PhD, Study Chair — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided